CLINICAL TRIAL: NCT03347903
Title: Prevalence and Clinical Characteristics of Patients With Jackhammer Esophagus and Symptoms of Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Ivan Kristo, Dr. med. univ., Medical University of Vienna
Other Study IDs: 1164/2017
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Esophageal Motility Disorders
Keywords: esophagus; motility
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastroesophageal reflux disease (GERD) is involved in the development of esophageal motility disorders like Jackhammer esophagus (JE), a novel hypercontractile condition that was associated with progression to achalasia and limited outcomes following surgical anti-reflux therapy.

This trial was designed to assess the prevalence and characteristics of JE in patients with typical symptoms of GERD and responsiveness to PPI therapy.

DETAILED DESCRIPTION:
Jackhammer esophagus is a novel hypercontractile esophageal disorder. The investigators assess the prevalence and clinical characteristics of patients diagnosed with this disorder out of a collective of patients that are referred with symptoms of gastroesphageal reflux disease and respond to PPI. This is an observational trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms of gastroesophageal reflux disease and diagnosis of Jackhammer esophagus

Exclusion Criteria:

* patients not willing to participate data or undergo screening for gastroesophageal reflux disease

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients that are referred to our center undergo esophageal high-resolution manometry and ambulatory pH monitoring for screening of gastroesophageal reflux disease and motility disorders. We assess the data that are prospectively obtained. Patients do not have to undergo any interventions.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Jackhammer esophagus in patients referred with symptoms of gastroesophageal reflux disease | January 2014- May 2017
  All patients that are referred to our center with symptoms of gastroesophageal reflux disease routinely undergo high-resolution manometry. We assess how many patients are diagnosed with Jackhammer esophagus

SECONDARY OUTCOMES:
Symptom perception | January 2014- May 2017
  We assess which symptoms are perceived by the patients diagnosed with Jackhammer esophagus. All data are observed during an interview at the high-resolution manometry
Prevalence of gastroesophageal reflux disease in patients with Jackhammer esophagus | Januar 2014- May 2017
  All patients that are referred to our center are evaluated for gastroesophageal reflux disease. We assess the prevalence of gastroesophageal reflux disease in patients with Jackhammer esophagus diagnosed by ambulatory pH monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Schoppmann, MD, Principal Investigator — Vice Chair of Department of General Surgery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kristo I, Schwameis K, Maschke S, Kainz A, Rieder E, Paireder M, Jomrich G, Schoppmann SF. Phenotypes of Jackhammer esophagus in patients with typical symptoms of gastroesophageal reflux disease responsive to proton pump inhibitors. Sci Rep. 2018 Jul 2;8(1):9949. doi: 10.1038/s41598-018-27756-9. PMID 29967357